CLINICAL TRIAL: NCT01455909
Title: A Phase 3, Randomized, Active Comparator, Double-Blind, Multi-Center Study to Compare the Efficacy, Safety and Tolerability of ITCA 650 to Sitagliptin as Add-on Therapy to Metformin in Patients With Type 2 Diabetes
Brief Title: A Study to Evaluate ITCA 650 Compared to Sitagliptin for the Treatment of Type 2 Diabetes
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Intarcia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITCA 650-CLP-110
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2012-12-25 (Estimated); Status verified 2012-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- ITCA 650 60 mcg/day (Experimental)
  Interventions: Drug: ITCA 650 60 mcg/day
- sitagliptin (Active Comparator): sitagliptin 100 mg/day
  Interventions: Drug: sitagliptin

INTERVENTIONS:
Drug: ITCA 650 60 mcg/day — exenatide in DUROS
  Arms: ITCA 650 60 mcg/day
Drug: sitagliptin — sitagliptin oral 100 mg/day
  Arms: sitagliptin

SUMMARY:
Phase 3 study to compare treatment with ITCA 650 to sitagliptin when added to metformin monotherapy in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c between 7.5%-10%
* on metformin monotherapy
* BMI between 25 & 45 kg/m2

Exclusion Criteria:

* taking thiazolidinedione, sulfonylurea, DPP-4, exenatide, alpha glucosidase inhibitors, meglitinides or insulin within last 3 months
* history of pancreatitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | 39 weeks
  39-week treatment period followed by 65-week extension period

CONTACTS AND LOCATIONS:
Locations (1):
- Intarcia Therapeutics, Inc, Hayward, California, United States